CLINICAL TRIAL: NCT06819527
Title: The Impact of Medication Reconciliation on Discrepancies and All-cause Readmission Among Hospitalized Patients With Chronic Kidney Disease: A Quasi-experimental Study
Brief Title: Medication Reconciliation in Hospitalized CKD Patients : A Quasi-Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Grant number: 20220257
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease(CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This was a quasi-experimental trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): interventional group, in which patients received a supplemented medication reconciliation service.
  Interventions: Other: Medication reconciliation service
- Retrospective control group in which patients received the usual care (No Intervention): A retrospective control group in which patients received the usual care that may or may not include medication reconciliation

INTERVENTIONS:
Other: Medication reconciliation service — Patients in the interventional group received medication reconciliation at admission and discharge in addition to continuous medication review during their admissions.
  Arms: Intervention group

SUMMARY:
This study aimed to evaluate the impact of combining medication reconciliation with medication review on reducing medication discrepancies at discharge and all-cause readmissions among CKD patients, in comparison to a retrospective control group that received usual care, which may or may not have included medication reconciliation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) admitted patients with CKD (stages 2-5 ), who were using at least three chronic medicines at home, and were hospitalized for at least 48 hours.

Exclusion Criteria:

* Patients with kidney transplantation .
* Patients who have difficulties in responding to interviews and did not have family member or caregiver on behave.
* Patients who refused to provide a written informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
all-cause 90-day readmission | 90 days after discharge
  The primary outcome in this study was the likelihood of all-cause 90-day readmission as extracted from medical records for both study groups

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah University Hospital and Princess Basma Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
The data generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Abu Farha R, Yousef A, Gharaibeh L, Alkhalaileh W, Mukattash T, Alefishat E. Medication discrepancies among hospitalized patients with hypertension: assessment of prevalence and risk factors. BMC Health Serv Res. 2021 Dec 14;21(1):1338. doi: 10.1186/s12913-021-07349-5. PMID 34903221